CLINICAL TRIAL: NCT04163627
Title: Epidemiology of Technical Procedures for the Treatment of Hepatocellular Carcinoma: Country-wide Trends From 2009 to 2019
Brief Title: Changing Trends in HCC Procedures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0505
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Hepatocellular Carcinoma
Keywords: Technical procedure for treatment of HCC: either liver transplantation, liver resection, thermal ablation, chemoembolization, or radioembolization; Chronic liver diseases; Interventional Radiology; Liver surgery
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In France, as in most countries, the incidence of primary liver cancer has increased significantly since the 1980s. In the United States, a study estimating cancer incidence and mortality rates in the coming years predicts that primary liver cancer will become the 3rd leading cause of cancer death from 2030 onwards, behind lung and pancreatic cancer, but ahead of colorectal cancer. This increase in incidence could be explained on the one hand by an increase in the incidence of chronic liver diseases, particularly those related to alcohol and metabolic steatopathies in the West, and on the other hand by improved management of the consequences of cirrhotic disease, which in turn increases the time needed for hepatocellular carcinoma (HCC) to form and develop. The management of a patient with hepatocellular carcinoma is complex because of the underlying cirrhotic disease, which hinders the development of many therapies. Thus, the patient's prognosis depends as much on the tumour extension as on the severity of the underlying chronic liver disease, and the choice of appropriate treatment is based on optimizing the balance between maximum antitumor efficacy and limited liver toxicity.

It is in this context that minimally invasive technical acts, whether local or local-regional, have developed significantly in recent years. Percutaneous tumor destruction techniques have become highly diversified with the development of microwave ablatherm, multipolar radiofrequency, or irreversible electroporation. For intra-arterial treatments, hepatic arterial chemoembolization remains the reference treatment for BCLC B stages. Alongside it, Yttrium 90 radio-embolization is booming, although its precise place remains to be defined in the therapeutic arsenal. Surgical techniques have also progressed, with the development of laparoscopic resections and improved liver transplant management. Finally, external radiotherapy is a recourse solution that can make it possible to propose a therapeutic solution in selected patients.

This multidisciplinary management of the HCC is in constant evolution and improvement, which justifies regularly carrying out an inventory of the frequency of these various technical acts at the national level. The objective of our study is to analyze the evolution, over the last 10 years and at a national level, of the various technical procedures available in the HCC therapeutic arsenal based on data from the french national PMSI database.

DETAILED DESCRIPTION:
Design Observational retrospective epidemiological nationwide cohort

Data source Data will be obtained from the French Programme for the Medicalisation of Information Systems (PMSI) database, which contains all discharge abstracts from all hospitals nationwide. The PMSI includes data on all hospital activities, whether acute (Medecine chirurgiae Obstetrique [MCO]), chronic (Soins de Suite et de Réadaptation [SSR]), or home-care (Hospitalization à Domicile [HAD]). Discharge abstracts include information on the patient's demographics, principal and associated diagnosis codes according to the tenth revision of the International Classification of Diseases (ICD-10) [10], procedure codes, mode of hospitalization (elective, emergency, or hospital transfer), mode of discharge (home, hospital transfer, death; the latter was used to compute survival), duration of hospital stay, patient's home address, and hospital identification code. In addition, each patient has an anonymous alphanumerical identifier that enables all hospital admissions throughout the country to be traced. The databases will be provided for the calendar years 2009 to 2018 included.

Data extraction

* date: 01/01/2009 to 31/12/2018
* ICD-10 diagnostic code: C22.0 (liver cell carcinoma - HCC or hepatoma) and C22.9 (malignant neoplasm of liver, unspecified)
* Patient: age, gender, co-morbidities, postal code
* Cause of chronic liver disease, presence of cirrhosis and severity
* 1st diagnosis of HCC or recurrence
* Hospital of care, status and postal code
* Number and type of therapeutic procedures performed per year (each procedure will be counted according to whether it is the first treatment of HCC or the treatment of a recurrence):

  * Liver transplantation
  * Destruction of hepatic tumor by radiofrequency, percutaneous
  * Destruction of hepatic tumor by radiofrequency, intraoperatively
  * Hepatectomy and liver resection:
  * Preoperative portal embolization
  * Liver arterial chemo-embolization:
  * Yttrium 90 Radio Embolization
* Survival from diagnosis and 1st treatment

The expected results of this study are of major importance. On the one hand, this study will provide an overview of the current situation regarding the management of HCC at a national level, by analysing the evolutionary trends of the various therapeutic solutions. The analysis of the geographical variability of care that may exist between different health structures at different levels of expertise, but also at regional or departmental level, is of major importance in order to detect and explain possible differences in terms of prognosis. These data may be of great interest to health authorities or to potential future investigators who will be committed to conducting new prospective projects based on solid and up-to-date data.

ELIGIBILITY:
Inclusion criteria:

An individual must fulfill all of the following criteria in order to be eligible for study enrollment:

* Aged above 18 years
* ICD-10 diagnostic code: C22.0 (liver cell carcinoma - HCC or hepatoma) and C22.9 (malignant neoplasm of liver, unspecified)
* Having had at least one technical procedure for management of an HCC
* Date of procedure: 01/01/2009 to 31/12/2018

Exclusion criteria:

* Age under 18
* Histological type different of HCC
* Systemic/oral or palliative treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with hepatocellular carcinoma with a technical procedure for the treatment of HCC: liver transplantation, liver resection, thermal ablation, chemoembolization or radioembolization
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-11-30 (Actual); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-03-25 (Estimated)

PRIMARY OUTCOMES:
Technical procedures evolutiveness | 1 day
  Quantify at the national level the progression from 2009 to 2019 in the number of procedures performed as part of the treatment of HCC, divided into percutaneous or intraoperative tumour destruction, chemo-embolisation, radio-embolisation, liver surgery and liver transplantation.

SECONDARY OUTCOMES:
Regional disparities | 1 day
  look for possible regional disparities according to prognosis and access to innovative care

CONTACTS AND LOCATIONS:
Overall Officials: BORIS GUIU, PU-PH, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC

REFERENCES:
- [Derived] Cassinotto C, Nogue E, Morell M, Panaro F, Molinari N, Guiu B. Changing trends in hepatocellular carcinoma management: Results from a nationwide database in the last decade. Eur J Cancer. 2021 Mar;146:48-55. doi: 10.1016/j.ejca.2021.01.009. Epub 2021 Feb 11. PMID 33582392